CLINICAL TRIAL: NCT00679861
Title: Different Types of Proactive Smoking Interventions for General Medical Practices: An Implementation Study
Brief Title: Smoking Interventions in General Medical Practices
Acronym: PRO GP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medicine Greifswald (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Research Foundation (Other)
Responsible Party: Christian Meyer (principal Investigator), Sabina Ulbricht (co-investigator), Ulrich John (study director), University of Greifswald, Institute of Epidemiology and Social Medicine
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: E2_P4, 01EB0420
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2008-05-19 (Estimated); Status verified 2008-05

CONDITIONS: Tobacco Smoking; Nicotine Dependence
Keywords: primary medical care; computer expert system; motivational interviewing; health behavior change counselling; stages of change
MeSH Terms: conditions — Tobacco Smoking; Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3 (Experimental): A practitioner delivered counselling and an expert system intervention is implemented in practices allocated to this arm
  Interventions: Behavioral: Counselling Intervention; Behavioral: Expert-system intervention
- 1 (Experimental): A practitioner delivered counselling intervention was implemented in practices allocated to this arm
  Interventions: Behavioral: Counselling Intervention
- 2 (Experimental): A computer expert system intervention was implemented in practices allocated to this arm
  Interventions: Behavioral: Expert-system intervention

INTERVENTIONS:
Behavioral: Counselling Intervention — A personal counselling by the residing practitioner of up to 10 minutes. A follow-up counselling is included for the next regular patient consultation
  Arms: 1; 3
Behavioral: Expert-system intervention — Counselling letter of three to four pages will be generated by an expert-system base on the assessment of the patient. A second and third letter will be generated at follow-up consultations.
  Arms: 2; 3

SUMMARY:
Primary care physicians can play an important role in reducing tobacco smoking in the population. The general practice is a suitable setting for implementing proactive smoking interventions, because a large proportion of the population can be regularly reached in a favorable psychological state. Further, a trustful interpersonal relationship between the practitioners and their patients is supposed to increase the susceptibility to preventive measures. However, currently general practitioners are not capitalizing this advantage although evidence based treatments are available, which are effective and cost-effective. Outreach programs combining educational and practice-based measures have been found to be effective in engaging practitioners in screening and in giving advice. Computer expert-system and brief counseling interventions, which are based on the Transtheo-retical Model of behavior change (TTM), are promising approaches for the entire population of practitioners and smoking patients. For large scale implementation, data are needed about the degree of integration in every day routine clinical practice that could be achieved by implementing such interventions. Objectives: Evaluating different strategies for the implementation of proactive smoking interventions in general practices. Methods: In a randomized controlled trial, 150 randomly selected general practices of a defined German region will be included. The procedure comprises the implementation of 1) an on-site computer expert-system intervention, 2) a counseling intervention provided by the practitioner, or 3) the computer expert-system plus the counseling intervention. During an implementation phase of one month, two on site training sessions and support by phone will be provided. Routine use of the interventions will be monitored for the following 6 months. Main outcome measures are the number and rate of identified and treated smokers. A follow-up assessment will be realized 12 months after practice attendance to determine the smoking status of the treated smokers.

ELIGIBILITY:
Inclusion Criteria:

* Practices with regular office hours
* Practices predominantly providing primary medical care for adults
* Patients with age 18 and older
* Patients with sufficient German language and cognitive capabilities to complete assessment
* Patients smoking within the preceding six month

Exclusion Criteria:

* Practices planing closure within the next 12 months
* Practices opening less than 12 months ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3215 (Estimated)
Dates: Start 2004-10; Primary Completion 2008-08 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Number of treated Patients by practice within study period | 7 months
Point prevalence smoking abstinence of treated patients | 24 hours, 7 days, 4 weeks, 6 months preceeding the 12 months follow-up assessment

SECONDARY OUTCOMES:
Participation rate of practices | within recruitment phase
Quit and cut down attempts of patients | 12 months
number of cigarettes smoked per day | 4 weeks preceeding follow-up
Stages of change progress | at 12 month follow-up compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyer, Dr., Principal Investigator — University of Greifswald; Ulrich John, Prof. Dr., Study Director — University of Greifswald